CLINICAL TRIAL: NCT06346041
Title: A Phase I Study of Evaluating the Safety and Efficacy of Intravenous IDOV-SAFETM in Patients With Advanced Solid Tumors
Brief Title: Safety and Efficacy of Intravenous IDOV-SAFETM in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HJG-IDOV-SAFE-LYSW
Record Dates: First submitted 2024-03-12; First posted 2024-04-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic Virus injection(IDOV-SAFETM) (Experimental): Intravenous administration of IDOV-SAFETM as single agent for patients with advanced solid tumors.
  Dose cohorts: 1x10^9 pfu、3x10^9 pfu、1x10^10 pfu and 3x10^10 pfu
  Interventions: Biological: Oncolytic Virus injection(IDOV-SAFETM)

INTERVENTIONS:
Biological: Oncolytic Virus injection(IDOV-SAFETM) — Administered by intravenous injection as single agent.

SUMMARY:
This is an open-label, dose escalation, phase I study to evaluate safety tolerability, MTD or MFD, pharmacokinetic profile, immunogenicity, and pharmacodynamic profile of IDOV-SAFETM in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study is a single agent dose escalation which will use an accelerated and "3+3" design to evaluate escalating doses of IDOV-SAFETM.Total enrollment will depend on the toxicities and/or activity observed, with approximately 13-19 evaluable participants enrolled. A Dose-Limiting Toxicity (DLT) observation period of 3weeks was established before the entry of the first patient at the next dose level. After all subjects in the current dose group have completed the DLT observation period, the administration of the next dose group can only be started if the condition of dose escalation is met.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign a written informed consent;
* Male and female, ≥18 years old and ≤75 years old;
* Histologically or cytologically confirmed advanced malignant solid tumors that do not respond to standard treatment (disease progression or treatment intolerance after treatment) or currently lack effective standard treatment (including but not limited to advanced MSS colorectal cancer);
* ECOG physical status score 0~1;
* Expected survival ≥3 months;
* At least one evaluable lesion according to the solid tumor response criteria (RECIST version 1.1). Note: If the only evaluable disease site has previously received radiation therapy, it can be considered an evaluable lesion after determining disease progression;
* Major organ and bone marrow functions meet the following criteria within 7 days prior to initial dosing:

  1. Blood routine: neutrophils ≥1.5×109/L, platelets > 100×109/L, hemoglobin ≥90g/L(no blood transfusion, no supportive treatment with G-CSF and other drugs within 2 weeks before screening);
  2. Liver function: General patients: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)≤3× upper limit of normal; Total bilirubin ≤1.5× upper limit of normal value; Patients with liver metastasis: ALT and/or AST ≤5× upper limit of normal;
  3. Renal function: serum creatinine (Cr)≤1.5× upper limit of normal value or creatinine clearance CCr≥60ml/min(using Cockcroft-Gault formula: The Ccr (ml/min) = [(140 - age) * weight kg * F] / [serum creatinine (mg/dl) x 72] (F = 1 male, the female F = 0.85).
  4. Coagulation function: prothrombin time (PT)≤ 1.5×ULN or International Normalized ratio (INR)≤ 1.5×ULN, and activated partial thromboplastin time (APTT)≤ 1.5×ULN;
* The blood pregnancy results of fertile female subjects within 7 days prior to the first dosing must be negative. Female subjects were willing to use highly effective contraception during the trial and for at least 90 days after the last dose of the trial drug. Male subjects were willing to use highly effective contraception during the trial and for at least 90 days after the last dose of the trial drug.

Exclusion Criteria:

* Severe systemic reactions or side effects due to prior smallpox vaccination;
* Patients with known to be allergic to the test drug or its excipients;
* Patients with a history of other tumors within 5 years prior to screening, excluding effectively resected cervical carcinoma in situ, low-risk gastrointestinal stromal tumor, breast cancer, cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and papillary thyroid carcinoma;
* Patients with untreated symptomatic central nervous system metastases (CNS) who meet one of the following criteria can be enrolled:

  1. CNS metastasis is asymptomatic and does not require treatment;
  2. The CNS metastases have been treated, neurological symptoms have returned to baseline (except for treatment-related residual signs or symptoms), glucocorticoids have been discontinued for at least 2 weeks prior to randomization, and imaging studies within 28 days prior to randomization suggest that the CNS lesions are radiographically stable.
* Pial metastasis;
* Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* Previous acceptance of oncolytic viruses, stem cells or gene therapy products;
* Patients with received systemic antitumor therapy, including but not limited to chemotherapy, endocrine therapy, and immunotherapy, within 4 weeks before the first dose; Oral small-molecule targeted drugs are administered 2 weeks before the first dose or within 5 half-lives of the drug (whichever is longer); Palliative radiotherapy within 14 days before the first dose; Participated in clinical trials of other antitumor drugs within 4 weeks; Received any Chinese herbal medicine or proprietary Chinese medicine for any anti-tumor indication within 2 weeks prior to initial administration;
* The adverse reactions of previous anti-tumor therapy have not returned to CTCAE 5.0 grade evaluation ≤ Class 1 (except toxicity judged by the investigator to have no safety risk);
* Patients with received surgery or interventional treatment (excluding tumor biopsy, puncture, etc.) or unhealed wounds, ulcers or fractures within 4 weeks prior to the first dose;
* Patients with a history of severe cardiovascular and cerebrovascular disease, including but not limited to: congestive heart failure ≥ Class II of the New York Heart Association (NYHA); Left ventricular ejection fraction (LVEF)<50%; QT interval (QTcF)>470ms as corrected by the Fridericia method or prolonged QT interval syndrome; Acute coronary syndrome, aortic dissection, severe arrhythmia, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first treatment; Hypertension poorly controlled by standard treatment (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
* Patients with a history of exfoliated skin that requires systemic treatment (such as eczema or ectopic dermatitis);
* Active hepatitis B (HbsAg positive, HBV DNA test value greater than the upper limit of normal); Active hepatitis C (those with positive anti-HCV antibodies are further tested positive for HCV RNA); A known history of immunodeficiency virus (HIV) disease or a positive HIV antibody test;
* Subject with an active infection or developed an unexplained fever > 38.5 ° C during screening or prior to initial administration;
* There is evidence of clinically significant immunodeficiency, such as a primary immunodeficiency state, such as severe combined immunodeficiency disease (SCID); Co-opportunistic infection;
* At the time of screening, patients with active autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc., or with a history of autoimmune diseases that may recur, except for the following conditions: (1)Type 1 diabetes; (2)Hypothyroidism (if controlled with hormone replacement therapy alone); (3)Controlled celiac disease; (4)Skin diseases that do not require systemic treatment;(5) Any other disease that will not recur in the absence of an external trigger;
* Subject with an active infection or developed an unexplained fever > 38.5 ° C during screening or prior to initial administration;are receiving long-term systemic steroid (prednisone >10mg/ day or equivalent dose of the same drug) or any other form of immunosuppressant therapy within 14 days prior to initial treatment; Treatment with topical, ocular, intra-articular, intranasal, and inhalation corticosteroids is excluded; Short-term use of corticosteroids (≤10mg equivalent dose of prednisone) for preventive treatment (e.g. prevention of contrast agent allergy);
* Patients with received allogeneic tissue or solid organ transplantation;
* Other diseases or abnormalities assessed by the investigator as unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Within day 21 after administration
  Dose-limiting toxicity is defined as an adverse event that is considered to be drug-related and meets one of the Protocol definitions
Incidence of adverse events and severe adverse events | Within day 85 after administration
  Graded according to the NCI CTCAE version 5.0
MTD/MFD | Within day 21 after administration
  To explore the maximum tolerated dose (MTD) or maximum administration dose (MFD) of IDOV-SAFETM in patients with advanced solid tumors.

SECONDARY OUTCOMES:
The Pharmacokinetics characteristics of IDOV-SAFETM((biological distribution and viral expulsion)) | Up to 2 days
  1. The level of (non-essential) viral DNA in tumor tissue;
  2. Levels of viral DNA in blood, saliva and urine
Immunogenicity of IDOV-SAFETM | Up to 85 days
  Neutralizing antibody titer
ORR | Every 6 weeks (±7 days) after initial administration and every 12 weeks (±7 days) after 1 year
  The sum of the proportion of subjects with CR or PR
DCR | Every 6 weeks (±7 days) after initial administration and every 12 weeks (±7 days) after 1 year
  The sum of the proportion of subjects with CR 、PR or SD
DOR | Every 6 weeks (±7 days) after initial administration and every 12 weeks (±7 days) after 1 year
  The time between the start of the first assessment of the tumor as CR or PR and the second assessment as PD(Progressive Disease) or death from any cause
PFS | Every 6 weeks (±7 days) after initial administration and every 12 weeks (±7 days) after 1 year
  The time, measured in days, from the date of first treatment to disease progression or death from any cause. Disease progression and death were measured in terms of preoccurrence. Progression included radiographic progression or clinical progression as assessed by the investigator.
OS | Up to death
  The time from the date of first treatment to death from any cause, measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No